CLINICAL TRIAL: NCT06552780
Title: High Intensity Laser Versus Ischemic Compression on Myofascial Trigger Points in the Upper Trapezius
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa mohamed abdelfatah elrefaey, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012\005287
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
Keywords: "myofascial pain syndrome" "trigger points" "high intensity laser " "ischemic compression"
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation; Ultrasonic Therapy; Lasers; Acupressure

STUDY DESIGN:
Intervention Model Description: Treatment
Who Masked: Participant
Masking Description: participants will be divided into three groups of equal number group A , group B ,and group C
  ,the randomization will be performed by computerized randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high intensity laser , TENs and ultrasound and isometric exercise (Experimental): Group A ( study group )will receive high intensity laser ,TENs , ultrasound therapy , and isometric exercise.
  Interventions: Device: TENs , ultrasound therapy
- ischemic compression ,TENs , ultrasound and isometric exercise (Experimental): Group B ( study group) will receive ischemic compression ,TENs and ultrasound therapy and isometric exercise.
  Interventions: Device: TENs , ultrasound therapy
- TENs , ultrasound and isometric exercise (Experimental): Group C (control group ) will receive TENs and ultrasound therapy and isometric exercise only.
  Interventions: Device: TENs , ultrasound therapy

INTERVENTIONS:
Device: TENs , ultrasound therapy — effect of high intensity laser versus ischemic compression on myofascial trigger points in the upper trapezius
  Other Names: high intensity (power) laser, ischemic compression; TENs , ultrasound therapy , isometric exercise and stretching exercise.

SUMMARY:
TO Investigate the effect of high intensity laser versus ischemic compression on myofascial trigger points on neck pain, cervical range of motion,pressure pain thershold and cervical disability and to show that the more effectivness therapy will provide significant clinical value

DETAILED DESCRIPTION:
Randomized controlled Trial , participants will be assigned into three groups (study group A ,study group B and study group c ) Subject selection will be 63 subjects , 21 subjects in each group with trigger points in the upper trapezius.

Groups

ELIGIBILITY:
Inclusion Criteria:

* The age of patients range from 20 to 50 years .
* patient Body mass index starting from 19 to 25 kg\m.
* presence of myofascial trigger points in the shortened upper trapezius muscle evaluated .

Exclusion Criteria:

* patients with fibromyalgia syndrome.
* cancer or tumor or any type diagnosed .
* patients with disc herniation or spinal canal stenosis.
* pregnancy -
* patients diagnosed with epilepsy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
cervical range of motion (CROM) | 30 seconds
  All the cervical active movements will be measured by cervical range of motion device (CROM) especially in cervical flexion ,extension and medial and lateral rotation.one tester will document the results.
  cervical range of motion (cROM) will be measured by using Electronic CROM Goniometer in all ranges.

SECONDARY OUTCOMES:
cervical pain | one minute
  Cervical pain will be measured by Cervical range of motion device (CROM) .The patient will actively perform cervical movements in flexion ,extension and medial and lateral rotation then one tester will document the results as VAS will be used to measure pain levels .The VAS is a 10_cm line divided into 10 equal sections , with 10 expressing "unbearable pain " and 0 indicating no pain .each patient will be asked to point on this line to their level of neck pain .as pain level decreases ,the patient state improves. Pain will be assessed before and after treatment.

OTHER OUTCOMES:
pressure pain threshold (PPT) | 10 seconds
  Pressure pain threshold (PPT) ,measured by Algometer is defined as the point at which painless stimulation such as pressure turns into a painful sensation,so that we will measure PPT for each patient before and after treatment by one tester as pressure Algometry is a method that objectively describes PPT

CONTACTS AND LOCATIONS:
Overall Officials: RAGIAA KAMEL, PROFFESOR DR, Principal Investigator — RAGIAA M KAMEL , PROF DR
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No